CLINICAL TRIAL: NCT03783845
Title: The Effects of Non -Surgical Periodontal Therapy on Glycemic Control and Periodontal Health in Diabetic Patients With Periodontitis (Randomized Controlled Clinical Trial)
Brief Title: The Effects of Periodontal Therapy on Glycemic Control in Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Yasser El Makaky, Associated professor, Taibah University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: periodontal therapy and HbA1c
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Chronic Periodontitis, Generalized
MeSH Terms: conditions — Chronic Periodontitis | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Metronidazole 400mg,three times daily for two weeks
  Amoxicillin 500mg,three times daily for two weeks.
  Interventions: Combination Product: amoxicillin 500mg and metronidazole 400mg
- control group (No Intervention): no intervention during study period

INTERVENTIONS:
Combination Product: amoxicillin 500mg and metronidazole 400mg — metronidazole 400mg and amoxicillin 500mg three times daily for two weeks
  Other Names: Amoxil and Flagyl
  Arms: test group

SUMMARY:
Is the non-surgical periodontal therapy can improve glycemic control in type 2 diabetic patients with chronic periodontitis?

DETAILED DESCRIPTION:
The aim of the present study was to monitor the clinical outcomes and the metabolic response of non-surgical periodontal therapy in patients with chronic periodontitis and uncontrolled type 2 diabetes.

Regarding clinical and metabolic parameters at baseline, no differences were displayed between two groups. However, at 3-months follow-up period the patients within a test group were demonstrated better clinical outcomes than patients in a control group

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of diabetes type 2 for more than five years Type 2 diabetes with HbA1c level from 7% to 9% at the last medical evaluation Diagnosis with chronic periodontitis

Exclusion Criteria:

Pregnancy

* Alcoholism and smoking
* Presence of any systemic disorders other than hypertension and diabetes
* Diabetic major complications

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
glycosylated haemoglobin (HbA1c) | 3 months
  Blood was taken from a peripheral vein to monitor HbA1c using high-performance liquid chromatography

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03783845/Prot_SAP_001.pdf